CLINICAL TRIAL: NCT00608218
Title: Ciclesonide for the Therapy of Asthma During the Cold Season.
Brief Title: Efficacy of Ciclesonide During the Cold Season in Patients Older Than 12 Years With Persistent Asthma
Acronym: ARTIST
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: Alves Artist 07/10
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Asthma; ciclesonide; inhaled steroids; Alvesco
MeSH Terms: conditions — Asthma | interventions — ciclesonide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Artist
  Interventions: Drug: Ciclesonide

INTERVENTIONS:
Drug: Ciclesonide — This is an observational study. Therefore, the physician decides about dosage according to individual needs.

SUMMARY:
The aim of the study is to evaluate the efficacy of ciclesonide in patients with persistent asthma over 3 months, especially in the cold season. Ciclesonide will be inhaled by a metered-dose inhaler. The study will provide further data on safety and tolerability of ciclesonide.

ELIGIBILITY:
Main inclusion criteria:

* History of persistent bronchial asthma

Main exclusion criteria:

* Hypersensitive to compounds of Alvesco
* Other criteria as defined in the Summary of Product Characteristics (Fachinformation Chapter 4.3)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
FEV1, symptom score assessment | within 3 months

SECONDARY OUTCOMES:
Handling of the metered-dose inhaler, safety and tolerability | within 3 months

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (122):
- Germany (122):
  - "Nycomed Deutschland GmbH", Adendorf
  - "Nycomed Deutschland GmbH", Arnstadt
  - "Nycomed Deutschland GmbH", Auerbach
  - "Nycomed Deutschland GmbH", Augsburg
  - "Nycomed Deutschland GmbH", Backnang
  - "Nycomed Deutschland GmbH", Bad Bramstedt
  - "Nycomed Deutschland GmbH", Bad Kreuznach
  - "Nycomed Deutschland GmbH", Bad Lippspringe
  - "Nycomed Deutschland GmbH", Bad Neuenahr-Ahrweiler
  - "Nycomed Deutschland GmbH", Bad Neustadt an der Saale
  - "Nycomed Deutschland GmbH", Bad Soden
  - "Nycomed Deutschland GmbH", Bad Tölz
  - "Nycomed Deutschland GmbH", Bautzen
  - "Nycomed Deutschland GmbH", Bergisch Gladbach
  - "Nycomed Deutschland GmbH", Berlin
  - "Nycomed Deutschland GmbH", Bietigheim-Bissingen
  - "Nycomed Deutschland GmbH", Braunschweig
  - "Nycomed Deutschland GmbH", Bredstedt
  - "Nycomed Deutschland GmbH", Breisach
  - "Nycomed Deutschland GmbH", Bremen
  - "Nycomed Deutschland GmbH", Bremerhaven
  - "Nycomed Deutschland GmbH", Bröckel
  - "Nycomed Deutschland GmbH", Bruchsal
  - "Nycomed Deutschland GmbH", Burgwedel
  - "Nycomed Deutschland GmbH", Castrop-Rauxel
  - "Nycomed Deutschland GmbH", Coburg
  - "Nycomed Deutschland GmbH", Cologne
  - "Nycomed Deutschland GmbH", Cottbus
  - "Nycomed Deutschland GmbH", Delitzsch
  - "Nycomed Deutschland GmbH", Dortmund
  - "Nycomed Deutschland GmbH", Dresden
  - "Nycomed Deutschland GmbH", Duisburg
  - "Nycomed Deutschland GmbH", Düren
  - "Nycomed Deutschland GmbH", Düsseldorf
  - "Nycomed Deutschland GmbH", Eisenach
  - "Nycomed Deutschland GmbH", Erfurt
  - "Nycomed Deutschland GmbH", Eschwege
  - "Nycomed Deutschland GmbH", Finsterwalde
  - "Nycomed Deutschland GmbH", Flensburg
  - "Nycomed Deutschland GmbH", Frankfurt
  - "Nycomed Deutschland GmbH", Freising
  - "Nycomed Deutschland GmbH", Friedrichshafen
  - "Nycomed Deutschland GmbH", Fürstenwalde
  - "Nycomed Deutschland GmbH", Garmisch-Partenkirchen
  - "Nycomed Deutschland GmbH", Gelsenkirchen
  - "Nycomed Deutschland GmbH", Gotha
  - "Nycomed Deutschland GmbH", Greiz
  - "Nycomed Deutschland GmbH", Hagen
  - "Nycomed Deutschland GmbH", Halle
  - "Nycomed Deutschland GmbH", Hamburg
  - "Nycomed Deutschland GmbH", Hanover
  - "Nycomed Deutschland GmbH", Hartha
  - "Nycomed Deutschland GmbH", Haßloch
  - "Nycomed Deutschland GmbH", Heidelberg
  - "Nycomed Deutschland GmbH", Heilbronn
  - "Nycomed Deutschland GmbH", Herne
  - "Nycomed Deutschland GmbH", Herten
  - "Nycomed Deutschland GmbH", Hoyerswerda
  - "Nycomed Deutschland GmbH", Höchstadt an der Aisch
  - "Nycomed Deutschland GmbH", Husum
  - "Nycomed Deutschland GmbH", Jettingen
  - "Nycomed Deutschland GmbH", Karlsruhe
  - "Nycomed Deutschland GmbH", Kiel
  - "Nycomed Deutschland GmbH", Koblenz
  - "Nycomed Deutschland GmbH", Konstanz
  - "Nycomed Deutschland GmbH", Laatzen
  - "Nycomed Deutschland GmbH", Leipzig
  - "Nycomed Deutschland GmbH", Limburg
  - "Nycomed Deutschland GmbH", Lohfelden
  - "Nycomed Deutschland GmbH", Mainz
  - "Nycomed Deutschland GmbH", Mannheim
  - "Nycomed Deutschland GmbH", Marburg
  - "Nycomed Deutschland GmbH", Markkleeberg
  - "Nycomed Deutschland GmbH", Menden
  - "Nycomed Deutschland GmbH", Minden
  - "Nycomed Deutschland GmbH", Moers
  - "Nycomed Deutschland GmbH", Mühlhausen
  - "Nycomed Deutschland GmbH", München
  - "Nycomed Deutschland GmbH", Neu Wulmstorf
  - "Nycomed Deutschland GmbH", Neubrandenburg
  - "Nycomed Deutschland GmbH", Neumarkt
  - "Nycomed Deutschland GmbH", Neuruppin
  - "Nycomed Deutschland GmbH", Neuss
  - "Nycomed Deutschland GmbH", Nordhausen
  - "Nycomed Deutschland GmbH", Oberursel
  - "Nycomed Deutschland GmbH", Offenburg
  - "Nycomed Deutschland GmbH", Osnabrück
  - "Nycomed Deutschland GmbH", Plauen
  - "Nycomed Deutschland GmbH", Radebeul
  - "Nycomed Deutschland GmbH", Rendsburg
  - "Nycomed Deutschland GmbH", Rosengarten
  - "Nycomed Deutschland GmbH", Rostock
  - "Nycomed Deutschland GmbH", Saalfeld
  - "Nycomed Deutschland GmbH", Saarbrücken
  - "Nycomed Deutschland GmbH", Saarlouis
  - "Nycomed Deutschland GmbH", Salzgitter
  - "Nycomed Deutschland GmbH", Schmölln
  - "Nycomed Deutschland GmbH", Schwalmtal
  - "Nycomed Deutschland GmbH", Schwarmstedt
  - "Nycomed Deutschland GmbH", Schwerin
  - "Nycomed Deutschland GmbH", Siegen
  - "Nycomed Deutschland GmbH", Sinsheim
  - "Nycomed Deutschland GmbH", Solingen
  - "Nycomed Deutschland GmbH", Sonneberg
  - "Nycomed Deutschland GmbH", Stadthagen
  - "Nycomed Deutschland GmbH", Starnberg
  - "Nycomed Deutschland GmbH", Steißlingen
  - "Nycomed Deutschland GmbH", Straelen
  - "Nycomed Deutschland GmbH", Stuttgart
  - "Nycomed Deutschland GmbH", Teterow
  - "Nycomed Deutschland GmbH", Teuchern
  - "Nycomed Deutschland GmbH", Uelzen
  - "Nycomed Deutschland GmbH", Ulm
  - "Nycomed Deutschland GmbH", Umkirch
  - "Nycomed Deutschland GmbH", Villingen-Schwenningen
  - "Nycomed Deutschland GmbH", Vilshofen
  - "Nycomed Deutschland GmbH", Wallertheim
  - "Nycomed Deutschland GmbH", Wilhelmshaven
  - "Nycomed Deutschland GmbH", Witten
  - "Nycomed Deutschland GmbH", Wörrstadt
  - "Nycomed Deutschland GmbH", Wörth
  - "Nycomed Deutschland GmbH", Würzburg